CLINICAL TRIAL: NCT01911676
Title: Translational Neuroscience Optimization of GlyT1 Inhibitor
Acronym: NCATS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1303011716; 4UH3TR000960-02 (NIH)
Record Dates: First submitted 2013-07-10; First posted 2013-07-30 (Estimated); Results first posted 2023-02-27 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Cognitive Impairments Associated With Schizophrenia
MeSH Terms: interventions — 1-methyl-1H-imidazole-4-carboxylic acid (3-chloro-4-fluoro-benzyl)-(3-methyl-3-aza-bicyclo(3.1.0) hex-6-ylmethyl)amide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PF-03463275 Active Dose #1 (Experimental): Active dose between 40mg
  Interventions: Drug: PF-03463275
- PF-03463275 Active Dose #2 (Experimental): Active dose between 60mg
  Interventions: Drug: PF-03463275
- Placebo (Placebo Comparator): Placebo- no active dose of PF-03463275.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-03463275
  Arms: PF-03463275 Active Dose #1; PF-03463275 Active Dose #2
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a Phase II, randomized, double-blind, placebo-controlled, cross-over POC study of stable patients with Schizophrenia or Schizoaffective disorder. The primary objective of this study is to test the efficacy of treatment with one of two does of a glycine transporter inhibitor (GlyT1I) combined with cognitive remediation to enhavce cognitive function. Subjects will be randomized to one of two doses of the glycine transporter inhibitor (GlyT1I) and placebo twice daily in addition to their antipsychotic medication for 2 treatment periods, each lasting a minimum of 5 weeks. Treatment periods will be separated by a washout period lasting approximately 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 1) Males or females 21 to 65 years of age (inclusive).
* 2) Diagnosis of Schizophrenia or Schizoaffective Disorder
* 3) Able to provide written informed consent.
* 4) Only CYP2D6 extensive metabolizers.

Exclusion Criteria:

* 1) No ongoing acute medical issues
* 2) Clinically significant ECG abnormality
* 3) Blood donation within eight weeks of the start of the study
* 4) Current treatment with Clozapine

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2013-08; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepak C D'Souza, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Connecticut Mental Health Center, New Haven, Connecticut
  - VA Connecticut Healthcare System, West Haven, Connecticut

REFERENCES:
- [Derived] Surti TS, Ranganathan M, Johannesen JK, Gueorguieva R, Deaso E, Kenney JG, Krystal JH, D'Souza DC. Randomized controlled trial of the glycine transporter 1 inhibitor PF-03463275 to enhance cognitive training and neuroplasticity in schizophrenia. Schizophr Res. 2023 Jun;256:36-43. doi: 10.1016/j.schres.2023.04.010. Epub 2023 May 2. PMID 37141764

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects will be randomized to one of two doses of PF-03463275 and placebo twice daily for 2 treatment periods each lasting approx 5 weeks. Treatment periods will be separated by a washout period lasting approx 3 weeks. The 4 possible study arms are as follows: A) Pd 1: Active dose 60mg PF-03463275 then Pd 2: Placebo B) Pd 1: Active dose 40mg PF-03463275 then Pd 2: Placebo C) Pd 1: Placebo then Pd 2: Active dose 60mg PF-03463275 D) Pd 1: Placebo 40mg PF-03463275 then Pd 2: Placebo.
Groups:
- PF-03463275 Active Dose #1: Subjects randomized to this arm will receive the following: Period 1) Active dose 60mg PF-03463275, then Period 2) Placebo.
- PF-03463275 Active Dose #2: Subjects randomized to this arm will receive the following: Period 1) Active dose 40mg PF-03463275, then Period 2) Placebo.
- Placebo, Active Dose #1: Subjects randomized to this arm will receive the following: Period 1) Placebo, then Period 2) Active Dose 60mg PF-03463275.
- Placebo, Active Dose #2: Subjects randomized to this arm will receive the following: Period 1) Placebo, then Period 2) Active Dose 40mg PF-03463275.
Period: Period 1 of Study
Arm/Group | PF-03463275 Active Dose #1 | PF-03463275 Active Dose #2 | Placebo, Active Dose #1 | Placebo, Active Dose #2
Started | 23 | 23 | 12 | 13
Completed | 17 | 21 | 11 | 10
Not Completed | 6 | 2 | 1 | 3
Not completed — Withdrawal by Subject | 4 | 2 | 1 | 2
Not completed — Physician Decision | 2 | 0 | 0 | 1
Period: Period 2 of Study
Arm/Group | PF-03463275 Active Dose #1 | PF-03463275 Active Dose #2 | Placebo, Active Dose #1 | Placebo, Active Dose #2
Started | 17 | 21 | 11 | 10
Completed | 15 | 21 | 11 | 8
Not Completed | 2 | 0 | 0 | 2
Not completed — Physician Decision | 2 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-03463275 Active Dose #1 | PF-03463275 Active Dose #2 | Placebo, Active Dose #1 | Placebo, Active Dose #2 | Total
Number analyzed (Participants) | 23 | 23 | 12 | 13 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 23 | 12 | 13 | 71
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 45.4 [25 to 61] | 49.6 [28 to 65] | 50.92 [27 to 64] | 39.77 [24 to 57] | 46.9 [24 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5 | 5 | 15
  Male | 21 | 20 | 7 | 8 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 3 | 2 | 9
  Not Hispanic or Latino | 21 | 21 | 9 | 11 | 62
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 16 | 14 | 5 | 6 | 41
  White | 6 | 7 | 7 | 5 | 25
  More than one race | 1 | 2 | 0 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB)
Description: To test the efficacy of PF-03463275 on cognitive test performance specifically, the MCCB composite score was used. The MCCB consists of 10 tests and provides standard scores and percentiles for each of seven cognitive domains and an overall composite score. Domains assessed include: speed of processing, attention/vigilance, working memory (verbal and visual), verbal learning, visual learning, reasoning and problem solving, and social cognition. The MCCB overall composite score is presented as a T-score. The range of T-scores is between 0 to 100 with a mean of 50 and standard deviation of 10. Higher scores indicate better overall cognitive functioning.
Time Frame: Change from baseline in cognitive measures at approximately 5 weeks. Mean scores were calculated per time point for each arm.
Population: The 3 arms that subjects can be randomized to are: A) Period 1: Active 60mg PF-03463275 then Period 2: Placebo; B) Period 1: Active 40mg PF-03463275 then Period 2: Placebo; C) Period 1: Placebo then Period 2: Active 60mg or 40mg PF-03463275. The following completed both period 1 and period 2 of the study: A) 15 subjects; B) 21 subjects; and C) 18 subjects (11 randomized to period 1-placebo/period 2-60mg PF-03463275; and 8 randomized to period 1-placebo/period 2-40mg PF-03463275).
Measure: Mean (Standard Deviation); unit: score on scale
Groups:
- PF-03463275 Active Dose #1: Period 1: Active dose 60mg PF-03463275
  Period 2: Placebo
- PF-03463275 Active Dose #2: Period 1: Active dose 40mg PF-03463275
  Period 2: Placebo
- Placebo, Active Dose #1: Period 1: Placebo
  Period 2: Active dose 60mg PF-03463275
- Placebo, Active Dose #2: Period 1: Placebo
  Period 2: Active dose 40mg PF-03463275
Arm/Group | PF-03463275 Active Dose #1 | PF-03463275 Active Dose #2 | Placebo, Active Dose #1 | Placebo, Active Dose #2
Number analyzed (Participants) | 15 | 21 | 11 | 8
score on scale
  Pre-Dose Period 1 | 28.15 (13.54) | 25.22 (13.86) | 31.71 (17.24) | 28.3 (17.7)
  Post-Dose Period 1 | 29.25 (12.38) | 26.33 (14.96) | 30.86 (17.45) | 30.11 (14.75)
  Pre-Dose Period 2 | 29.39 (12.68) | 27.11 (12.46) | 32.86 (18.52) | 31.8 (16.5)
  Post-Dose Period 2 | 31.84 (13.36) | 28.21 (11.49) | 34.29 (18.88) | 32.2 (16.01)

2. Secondary Outcome: Alteration in Symptom Domain Scores and Event Related Potentials (ERPs) With PF-03463275
Description: To determine whether PF-03463275 impacts symptom domain scores and visual event related potentials (ERPs), analogous to long-term potentiation (LTP) with PF-03463275 treatment. A more positive value reflects a better outcome - there is no established range to report. A Z-score of 0 indicates the mean score. A positive z-score indicates the mean is higher than average.
Time Frame: Change from Baseline at approximately 1 week
Population: Noncompleters and unusable data of completers led to differences between the total number of participants and the sample for this outcome measure.
Measure: Mean (Standard Error); unit: Mean LTP Standard (z) Score +1 SE
Groups:
- Placebo, Active Dose #1: Period 1: Placebo
  Period 2: Active dose 60mg
Arm/Group | PF-03463275 Active Dose #1 | PF-03463275 Active Dose #2 | Placebo, Active Dose #1 | Placebo, Active Dose #2
Number analyzed (Participants) | 14 | 18 | 9 | 6
Mean LTP Standard (z) Score +1 SE
  Pre-Dose Period 1 | -0.169 (0.221) | 0.084 (0.224) | -0.629 (0.267) | -0.111 (0.456)
  Post-Dose Period 1 | -0.544 (0.281) | -0.013 (0.188) | 0.228 (0.221) | 0.606 (0.300)
  Pre-Dose Period 2: number analyzed (Participants) | 12 | 16 | 9 | 6
  Pre-Dose Period 2 | -0.008 (0.323) | 0.473 (0.182) | -0.614 (0.398) | 0.127 (0.443)
  Post-Dose Period 2: number analyzed (Participants) | 12 | 16 | 9 | 6
  Post-Dose Period 2 | -0.129 (0.150) | 0.594 (0.316) | -0.674 (0.313) | 0.915 (0.421)

ADVERSE EVENTS:
Time Frame: Adverse events were captured from the time at which the participant signed consent throughout their completion in the study (follow up visit after the completion of period 2), over a time period of approximately 4 months.
Groups:
- PF-03463275 Active Dose #1: AEs while taking PF-03463275 Active Dose #1
- PF-03463275 Active Dose #2: AEs while taking PF-03463275 Active Dose #2
- Placebo: AEs while taking Placebo
- Washout: AEs while in the washout period (no medication)
Arm/Group | PF-03463275 Active Dose #1 | PF-03463275 Active Dose #2 | Placebo | Washout
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/33 | 0/63 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/34 | 2/33 | 0/63 | 0/59
Other Adverse Events (participants affected / at risk) | 13/34 | 13/33 | 9/63 | 7/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-03463275 Active Dose #1 (N=34) | PF-03463275 Active Dose #2 (N=33) | Placebo (N=63) | Washout (N=59)
Hospitalization from Intent to Overdose on Meds / Suicidal Ideation (Social circumstances) | 0 | 1 | 0 | 0
Hospitalization Due to Stroke (General disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-03463275 Active Dose #1 (N=34) | PF-03463275 Active Dose #2 (N=33) | Placebo (N=63) | Washout (N=59)
Increased Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Blurry Vision (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Sleep Disturbance (General disorders) | 0 (0) | 2 (2) | 4 (4) | 1 (1)
Hand Tremor (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lightheadedness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
High Blood Pressure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sprained Ankle (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foul Smelling Odor in Urine (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bell's Palsy (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (General disorders) | 3 (4) | 3 (3) | 2 (4) | 2 (2)
GI Discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness (General disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bruised Forearms (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated AST/ALT (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Knee Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry Cough (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower Back Strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hot Flashes (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Reduced Appetite (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Whiplash (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Trigeminal Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic Hypotension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Common Cold (General disorders) | 3 (3) | 1 (1) | 1 (1) | 5 (5)
Tooth Pulled (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Stomach Cramps/Discomfort (General disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Foot Injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Increased Sleep (General disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Nausea / Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
Laryngitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vasovagal Response (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dehydration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increase in Pain as a Result of Spinal Surgery Prior to Study (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal Ideation Due to Psychosocial Stressors (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Reduced Sleep (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Upper Respiratory Infection (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased Appetite (General disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Increase in Pre-Existing Headache (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive Cough / Chest Congestion (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Increase in Fibromyalgia Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye Sensitivity (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intermittent Blurred Vision (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Right Middle Finger) (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Low Mood (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Increased Urination (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Decreased Sleep (Associated with Pre-Existing Sleep Apnea) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased Discomfort Associated with Pre-Existing Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute Ear Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intermittent Dental Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gum Soreness (at site of tooth extraction) (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Throat Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sore Shoulder (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cold Symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contact Dermatitis on Forehead (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Stiffness (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Light Sensitivity (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip Pain (associated with pre-existing bone spur) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia in Right Lung (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus Congestion (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrist Drop / Radial Nerve Palsy (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Front Tooth Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-05-28): https://cdn.clinicaltrials.gov/large-docs/76/NCT01911676/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-28): https://cdn.clinicaltrials.gov/large-docs/76/NCT01911676/SAP_001.pdf
  • Informed Consent Form (2018-07-12): https://cdn.clinicaltrials.gov/large-docs/76/NCT01911676/ICF_002.pdf